CLINICAL TRIAL: NCT01259362
Title: Efeitos da Estimulacao Magnetica Transcrania de Repeticao ( EMTr) no Tratamento da Dependencia ao Uso de Cocaina
Brief Title: Effects of Repeated Transcranial Magnetic Stimulation (rTMS) on the Treatment of Cocaine Addicted Patients
Acronym: TMSCOCDEPEND
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Philip Leite Ribeiro, Department and Institute of Psychiatry, General Hospital University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLRIBEIRO1
Record Dates: First submitted 2010-12-10; First posted 2010-12-14 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-09

CONDITIONS: Cocaine Addiction; Treatment; Transcranial Magnetic Stimilation
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (Active Comparator): Cocaine addicted will receive a 20 day TMSr to right dorsolateral prefrontal cortex.
  Interventions: Procedure: Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimlation (Sham Comparator): cocaine addicted will receive a 20 day sham TMSr to right dorsolateral prefrontal cortex
  Interventions: Procedure: Transcranial Magnetic Stimulation

INTERVENTIONS:
Procedure: Transcranial Magnetic Stimulation — 5 Hz, 120 % motor threshold, intertrain interval 20s, number of pulses in train 50.
  Other Names: rTMS; Cocaine Addiction; Cocaine Addiction Treatment
  Arms: Transcranial Magnetic Stimulation
Procedure: Transcranial Magnetic Stimulation — Cocaine addicted will receive 20 sham TMSr
  Other Names: TMS; Cocaine Addiction; Sham Stimulation
  Arms: Transcranial Magnetic Stimlation

SUMMARY:
Cocaine addiction is a serious disease. Nowadays we still have no efficient method reducing craving and extending the abstinence period of this patients during treatment.

The aim of this study is to evaluate reduction if craving and other parameters related to addiction within this group of patients through a treatment with transcranial magnetic stimulation.

DETAILED DESCRIPTION:
Patients are going to submitted do a course of rTMS of one month, each session up to 15 minutes.

After the rTMS they are going to be offered cognitive therapy to prevent relapse.

The area stimulated is the dorso-lateral prefrontal cortex. This technique was employed in previous studies and the risks are insignificant.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18
* Maximum age of 40
* Diagnostic of Cocaine addiction
* Willingly participate the study

Exclusion Criteria:

* Metallic Cerebral Implant
* History of Severe Brain trauma or injury
* Organic Brain Disease
* Severe Somatic Disease
* History of other actual or past psychiatric diagnostics

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Minnesota Cocaine Craving Scale(MCCS) | 2 months
  Reduction on the scores of MCCS

SECONDARY OUTCOMES:
Barrat Impulsiveness Scale vers 11 ( BIS 11) | 2 months
  Reduction of scores of BIS 11.

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Ribeiro, MD, Principal Investigator — Post Graduate Student Department of Brain Stimulation - IPQ - HC FMUSP
Locations (1):
- Department and Institute of Psychiatry, General Hospital, University of Sao Paulo medical school, São Paulo, São Paulo, Brazil